CLINICAL TRIAL: NCT03808090
Title: Obesity and Endogenous Oxalate Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kyle D. Wood, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB130502007-OBE; 1K08DK115833-01A1 (NIH)
Record Dates: First submitted 2018-12-26; First posted 2019-01-17 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: oxalate; obesity; kidney stones
MeSH Terms: conditions — Obesity; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal Individuals (Experimental): Normal individuals: no prior history of kidney stones
  Interventions: Dietary Supplement: Normal Individuals

INTERVENTIONS:
Dietary Supplement: Normal Individuals — Controlled Dietary phase: Low oxalate fixed diet
  4 days of fixed normal calorie diet with low oxalate (< 60 mg/day), normal calcium (800-1200 mg/day)

SUMMARY:
The goal of this study is to determine if obesity is associated with increased endogenous oxalate synthesis as assessed by urinary oxalate excretion, which is a known risk factor for calcium oxalate kidney stones.

The study will recruit adult participants without history of kidney stones. Participants will

* Ingest fixed diets containing low amounts of oxalate for 4 days
* Collect 24-hr urine samples during the fixed diet

DETAILED DESCRIPTION:
In this study the investigators propose to measure the excretion of urinary oxalate on a fixed diet with controlled amounts of oxalate, in individuals of varying body sizes without history of kidney stones. The 24-hr urinary oxalate excretion on such a low-oxalate normal calcium fixed diet is determined to be an appropriate surrogate for endogenous oxalate synthesis.

Screening phase. The study will enroll 60 individuals without history of kidney stones (30 males/30 females) at the University of Alabama at Birmingham (UAB).

Screening will include blood complete metabolic profile, 24-hr urine specimens collected at home on self-selected diets and anthropometric measurements.

Dietary phase Participants will ingest a low-oxalate (<60 mg/day), normal calcium (1000 mg/day) fixed diet for 4 consecutive days, collect three 24-hr urines after 1 day of dietary equilibration and have a fasted blood draw on day 5.

ELIGIBILITY:
Inclusion Criteria

Age 19-70 yrs Body Mass Index > 18.5 kg/m2 Normal fasting serum electrolytes on comprehensive metabolic profile Willing to ingest fixed diets

Exclusion Criteria

Chronic Kidney Disease, estimated glomerular filtration rate < 60 ml/mn/1.73m2 Primary hyperoxaluria Liver, endocrine or renal diseases or any other condition that may influence the absorption, transport or urinary excretion of ions, which will compromise the interpretation of results, including: Cystic fibrosis, Cystinuria, Uric acid stone former, Nephrotic syndrome, Sarcoidosis, Renal tubular acidosis, Primary hyperparathyroidism, Neurogenic bladder, Urinary diversion Pregnancy or breast-feeding Incompatible dietary requirements with the study, food allergies or intolerance to any of the foods in study menus Active malignancy or treatment for malignancy within 12 months prior to screening Utilization of immunosuppressive medication Uncontrolled Hypertension or diabetes

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle D Wood, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: total study enrollment
Groups:
- Normal Individuals: Normal individuals: no prior history of kidney stones
  Normal Individuals: Controlled Dietary phase: Low oxalate fixed diet
  4 days of fixed eucaloric diet with low oxalate (< 60 mg/day), normal calcium (800-1200 mg/day)
Period: Overall Study
Arm/Group | Normal Individuals
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Normal Individuals
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 58
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29 (7)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Oxalate Excretion
Description: Mean Urinary oxalate excretion from three 24 hour urine collections on the fixed diet (mg/day)
Time Frame: 3 days on the fixed diet
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Normal Individuals
Number analyzed (Participants) | 58
mg/day | 24 (10)

2. Secondary Outcome: Urinary Glycolate Excretion
Description: mean of three 24-hr urinary glycolate collected on the fixed diet (mg/day)
Time Frame: 3 days on fixed diet
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Normal Individuals
Number analyzed (Participants) | 58
mg/day | 32 (14)

3. Secondary Outcome: Urinary Creatinine Excretion
Description: mean of there 24hr urinary creatinine excretion on the fixed diet ( g/day)
Time Frame: 3 days on the fixed diet
Measure: Mean (Standard Error); unit: g/day
Arm/Group | Normal Individuals
Number analyzed (Participants) | 58
g/day | 1.47 (0.58)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Normal Individuals
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03808090/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT03808090/ICF_001.pdf